CLINICAL TRIAL: NCT03519945
Title: A Phase 3, Multicenter, Open-Label Extension Study to Evaluate the Long Term Efficacy and Safety of Mirikizumab in Patients With Moderately to Severely Active Ulcerative Colitis LUCENT 3
Brief Title: A Study to Evaluate the Long-Term Efficacy and Safety of Mirikizumab in Participants With Moderately to Severely Active Ulcerative Colitis (LUCENT 3)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16596; I6T-MC-AMAP (Other: Eli Lilly and Company); 2017 004092 31 (EudraCT Number); 2023-507657-15-00 (Other: EUCTR)
Record Dates: First submitted 2018-05-07; First posted 2018-05-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirikizumab (Experimental): Mirikizumab administered subcutaneously (SC).
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered SC.
  Other Names: LY3074828

SUMMARY:
This study is designed to evaluate the long-term efficacy and safety of mirikizumab in participants with moderately to severely active ulcerative colitis (UC). The study will last up to 3 years. Participants who complete the 3-year study may continue to receive mirikizumab until it is (outside of this study) in their country or until they meet other discontinuation criteria.

ELIGIBILITY:
* Inclusion Criteria

  * Participants from Study AMAC (NCT02589665) or AMBG (NCT03524092) who have had at least one study drug administration and have not had early termination of study drug.
  * Female participants must agree to contraception requirements.
* Exclusion Criteria

  * Participants must not have developed a new condition, including cancer in the originator study.
  * Participants must not have any important infections including, but not limited to, hepatitis B, hepatitis C, HIV/AIDS, and active tuberculosis (TB) during either originator study
  * Participants may not have received surgery for UC in the originator study or are likely to require surgery for treatment of UC during the study.
  * Participants must not have developed adenomatous polyps during the originator study that have not been removed prior to the start of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1063 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants in Clinical Remission | Week 52
  Clinical remission based on the modified Mayo Score (MMS).

SECONDARY OUTCOMES:
Percentage of Participants in Endoscopic Remission | Week 52
  Endoscopic remission based on the MMS Endoscopic Subscore (ES).
Percentage of Participants in Corticosteroid-free Remission | Week 52
  Participants in corticosteroid-free remission.
Percentage of Participants with Histologic-Endoscopic Mucosal Remission at Week 52 | Week 52
  Endoscopic remission based on the MMS ES and histologic remission based on histologic disease activity index.
Health Related Quality of Life: Inflammatory Bowel Disease Questionnaire (IBDQ) Score | Baseline to Week 52
  Health Related Quality of Life based on IBDQ score.
UC Symptoms: Numeric Rating Score | Week 160
  UC symptoms based on numeric rating score.
Percentage of Participants Who are Hospitalized Due to UC | Baseline to Week 160
  Participants who are hospitalized due to UC.
Percentage of Participants Who Undergo UC Surgeries Including Colectomy | Baseline to Week 160
  Participants who undergo UC surgeries including colectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (352):
- United States (48):
  - Digestive Health Specialists, Dothan, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Valleywise Health Medical Center, Phoenix, Arizona
  - InSite Digestive Health Care, Arcadia, California
  - Care Access - Berkeley, Berkeley, California
  - Om Research LLC, Lancaster, California
  - California Medical Research Associates, Northridge, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Direct Helpers Research Center, Hialeah, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Clintheory Healthcare, Orlando, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Florida Medical Clinic LLC, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - NorthShore University HealthSystem - Evanston Hospital, Evanston, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - GI Alliance Research Baton Rouge, Baton Rouge, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Nola Research Works, LLC, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Medical Center - Columbus Center, Novi, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - MNGI Digestive Health - Plymouth Endoscopy Center & Clinic, Plymouth, Minnesota
  - Columbia University Medical Center, New York, New York
  - Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Carolina Digestive Diseases and Endoscopy Center, Greenville, North Carolina
  - Care Access - Youngstown, Poland, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Central Sooner Research - Oklahoma - Northwest 47th Street, Oklahoma City, Oklahoma
  - Care Access - Pottsville, Pottsville, Pennsylvania
  - Digestive Disease Associates, Wyomissing, Pennsylvania
  - Midwest Medical Care, Sioux Falls, South Dakota
  - GI Alliance, Garland, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Southern Star Research Institute, San Antonio, Texas
  - GI Alliance, Southlake, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Care Access-Ogden, Ogden, Utah
  - Care Access Research LLC - Salt Lake City, Salt Lake City, Utah
  - Carilion Clinic, Roanoke, Virginia
  - Washington Gastroenterology - Tacoma, Tacoma, Washington
- Argentina (5):
  - Mautalen Salud e Investigación, Buenos Aires
  - CER medical Institute, Quilmes
  - Fundacion Estudios Clinicos, Rosario
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman
  - C.I.C.E. 9 de Julio, San Miguel de Tucumán
- Australia (7):
  - Royal Adelaide Hospital, Adelaide
  - Box Hill Hospital, Box Hill
  - Mater Misericordiae Limited, Brisbane
  - Princess Alexandra Hospital, Brisbane
  - Coastal Digestive Health, Maroochydore
  - St Vincent's Hospital, Melbourne
  - The Royal Melbourne Hospital, Parkville
- Austria (3):
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Uniklinikum Salzburg, Salzburg
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (3):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier de Wallonie Picarde - Site Notre Dame, Tournai
- Canada (9):
  - CISSS de la Monteregie-Centre, Greenfield Park
  - Victoria Hospital, London
  - University Hospital - London Health Sciences Centre, London
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal
  - Montreal General Hospital, Montreal
  - Fraser Clinical Trials Inc, New Westminster
  - Vancouver General Hospital, Vancouver
  - GIRI GI Research Institute - Vancouver, Vancouver
  - PerCuro Clinical Research, Victoria
- China (33):
  - Xiangya Hospital Central South University, Changsha
  - Changzhou No.2 People's Hospital, Changzhou
  - West China Hospital of Sichuan University, Chengdu
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Hainan General Hospital, Haikou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - The Second Affiliated hospital of Zhejiang University school of medicine, Hangzhou
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Anhui Provincial Hospital, Hefei
  - Center-Jilin Center Hospital, Jilin
  - Shandong Provincial Hospital, Jinan
  - Qilu Hospital of Shandong University, Jinan
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - The First People's Hospital of Yunnan Province, Kunming
  - Liaocheng People's Hospital, Liaocheng
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The Second Afilliated Hospital of Hebei Medical University, Shijiazhuang
  - Taian City Central Hospital, Taian
  - The 2nd Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - ZhuZhou Central Hospital, Zhuzhou
- Czechia (9):
  - Vojenská Nemocnice Brno, Brno
  - Fakultni Nemocnice u sv. Anny v Brne, Brno
  - Hepato-Gastroenterologie HK, Hradec Králové
  - MUDr. Gregar, s.r.o., Olomouc
  - PreventaMed, Olomouc
  - A-Shine, Pilsen
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - MEDIENDO, Prague
  - ISCARE klinicke centrum, Prague
- Denmark (3):
  - Herlev and Gentofte Hospital, Copenhagen
  - Sjællands Universitetshospital Køge, Køge
  - Sygehusenheden Nyborg, Nyborg
- France (13):
  - CHU d'Amiens-Picardie - Hôpital Sud, Amiens
  - CHRU Troussau, Chambray-lès-Tours
  - Hopital Claude Huriez - CHU de Lille, Lille
  - Chu Saint Eloi, Montpellier
  - Centres Médico Chirurgicaux - Clinique Ambroise Paré, Neuilly-sur-Seine
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier de Pau, Pau
  - CHU Bordeaux Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord, Saint-Priest-en-Jarez
  - Nouvel Hôpital Civil (NHC), Strasbourg
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
- LLC ARENSIA Exploratory Medicine, Tbilisi, Georgia
- Germany (8):
  - Charite Universitätsmedizin Berlin Campus Benjamin Franklin, Berlin
  - Krankenhaus Waldfriede, Berlin
  - Städtisches Klinikum Brandenburg, Brandenburg
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle
  - Universitätsklinikum Halle, Halle
  - HaFCED e.K. - Hamburgisches Forschungsinstitut für chronisch entzündliche Darmerkrankungen, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Haus der Gesundheit, Ludwigshafen
- Hungary (8):
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház, Békéscsaba
  - Semmelweis University, Budapest
  - Eszak-budai Szent Janos Centrumkorhaz, Budapest
  - Petz Aladar Egyetemi Oktato Korhaz, Győr
  - Endomedix Diagnosztikai Központ - Miskolc, Miskolc
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - CLINFAN Szolgáltató Kft, Szekszárd
  - Jávorszky Ödön Kórház, Vác
- India (12):
  - Apollo Hospitals Ahmedabad, Ahmedabad
  - M S Ramaiah Medical College and Hospitals, Bangalore
  - Owaisi Hospital and Research Center, Hyderabad
  - SR Kalla Memorial Gastro & General Hospital, Jaipur
  - Dayanand Medical College and Hospital, Ludhiana
  - Midas Multispeciality Hospital Pvt.Ltd., Nagpur
  - Fortis Hospital, Noida
  - Grant Medical Foundation - Ruby Hall Clinic, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Gandhi Hospital, Secunderabad
  - Nirmal Hospital, Surat
  - Acharya Vinoba Bhave Rural Hospital, Wardha
- Beaumont Hospital, Dublin, Dublin, Ireland
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center, Tel Aviv
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (9):
  - Azienda Ospedaliera Mater Domini, Catanzaro
  - Ospedale San Martino, Genova
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Ospedale Di Circolo, Rho
  - Fondazione Policlinico Tor Vergata, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Ospedale Sandro Pertini, Rome
  - Humanitas, Rozzano
  - Ospedale Mauriziano, Torino
- Japan (44):
  - Asahikawa City Hospital, Asahikawa
  - Tokyo Medical and Dental University Hospital, Bunkyō
  - Juntendo University Hospital, Bunkyō City
  - Mitsui Memorial Hospital, Chiyoda-ku
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Chuo-ku, Sapporo-shi
  - Sai Gastroenterologist Proctology, Fujiidera
  - Fukuoka University Hospital, Fukuoka
  - Matsuaikai Matsuda Hospital, Hamamatsu
  - Mito Medical Center, Higashiibaraki
  - National Hospital Organization Hirosaki National Hospital, Hirosaki
  - Sameshima Hospital, Kagoshima
  - Ofuna Central Hospital, Kamakura
  - Kawasaki Municipal Hospital, Kawasaki
  - Kitakyushu Municipal Medical Center, Kitakyusyu-shi
  - Aoyama Clinic GI Endoscopy & IBD Center, Kobe
  - Showa University Koto Toyosu Hospital, Kōtoku
  - Kumagaya General Hospital, Kumagaya-shi
  - Hidaka Coloproctology Clinic, Kurume-shi
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Gunma University Hospital, Maebashi
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Nagaoka Chuo General Hospital, Nagaoka
  - Hyogo College of Medicine, Nishinomiya
  - Okayama University Hospital, Okayama
  - Infusion Clinic, Osaka
  - National Hospital Organization - Osaka National Hospital - Institute For Clinical Research, Osaka
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Saga-Ken Medical Center Koseikan, Saga
  - Tokitokai Tokito Clinic Coloproctology Center, Saitama
  - Toho University Sakura Medical Center, Sakura
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Takagi Clinic - Sendai, Sendai
  - Jichi Medical University Hospital, Shimotsuke
  - Center Hospital of the National Center for Global Health and Medicine, Shinjyuku-ku
  - Kagawa Prefectural Central Hospital, Takamatsu
  - National Hospital Organization Takasaki General Medical Centar, Takasaki
  - Tokyo Yamate Medical Center, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
  - Mie University Hospital, Tsu
  - Matsushima Hospital, Yokohama
  - Yokohama City University Medical Center, Yokohama
  - Showa University Northern Yokohama Hospital, Yokohama
- Latvia (3):
  - Digestive Diseases Center "Gastro", Riga
  - Pauls Stradins Clinical Univeristy Hospital, Riga
  - RIGA EAST UNIVERSITY HOSPITAL ,Oncology Centre of Latvia, Riga
- Lithuania (5):
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Viesoji Istaiga Klaipedos Miesto Poliklinika, Klaipėda
  - Republic Hospital of Klaipeda, Klaipėda
  - Respublikine Panevezio ligonine, Panevezys
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Malaysia (3):
  - Hospital Serdang, Kuala Selangor
  - Hospital Universiti Sains Malaysia, Kubang Kerian
  - University Malaya Medical Centre, Lembah Pantai
- Mexico (3):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Centro Para El Desarrollo de La Medicina Y de Asistencia Medica Especializada S.C., Culiacán
  - Sociedad de Metabolismo y Corazon, Veracruz
- Republican Clinical Hospital, Chisinau, Moldova
- Netherlands (4):
  - Amsterdam UMC, locatie VUmc, Amsterdam
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Ziekenhuis Bernhoven, Uden
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (24):
  - Promedica Dental Clinic, Będzin
  - Centrum Medyczne "Medis" Manermed, Bydgoszcz
  - Centrum Medyczne Pratia Bydgoszcz, Bydgoszcz
  - Szpital Miejski im. Jana Pawła II w Elblagu, Elblag
  - All-Medicus, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Topolowa Medicenter, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - ZOZ Gastromed, Lublin
  - Medicenter Nowy Targ, Nowy Targ
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Centrum Medyczne LUX MED - Rzeszow, Rzeszów
  - Endoskopia Sp. z.o.o., Sopot
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - SONOMED Centrum Medyczne, Szczecin
  - Gastromed, Torun
  - NZOZ Formed, Wadowice
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Vivamed Sp. z o.o., Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Planetmed, Wroclaw
  - LexMedica, Wroclaw
  - ETG Zamość, Zamość
- Romania (5):
  - SC Memorial Healthcare International SRL, Bucharest
  - Monza - Ares, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - CCBR Clinical Research, Bucharest
  - Spitalul Pelican, Oradea
- Russia (19):
  - Poliklinika Agmu "Konsul'tativno-Diagnosticheskiy Tsentr", Barnaul
  - Scientific Centre of Reconstructive and Restorative Surgery, Irkutsk
  - Alliance Biomedical URAL Group, Izhevsk
  - Kazan State Medical University, Kazan'
  - SIH Kemerovo Regional Clinical Hosptial, Kemerovo
  - Nizhny Novgorod Regional Hospital N.A. Semashko, Nizhny Novgorod
  - Medical Center SibNovoMed, Novosibirsk
  - Research Institute of Physiology and Fundamental Medicine, Novosibirsk
  - Ultramed, Omsk
  - Karelia Republican Hospital V.A. Baranova, Petrozavodsk
  - Rostov State Medical University, Rostov-on-Don
  - North-Western State Medical University named after I.I.Mechnikov, Saint Petersburg
  - City Mariinskaya Hospital, Saint Petersburg
  - Scientific research center ECO-security, Saint Petersburg
  - First Pavlov State Medical University of Saint Petersburg, Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution City Clinical Hospital No.31, Saint Petersburg
  - Stavropol State Medical University, Stavropol
  - SHI of Yaroslavl Region Clinical Hospital #8, Yaroslavl
  - LLC MA New Hospital, Yekaterinburg
- Serbia (6):
  - Clinical Hospital Center Zvezdara, Belgrade
  - University Medical Center "Bezanijska kosa", Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Regional Hospital Dr Radivoj Simonovic Sombor, Sombor
  - Sremska Mitrovica Health Centre, Sremska Mitrovica
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (5):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica
  - Cliniq s.r.o., Bratislava
  - KM Management, Nitra
  - Gastro, Prešov
  - Endomed, s.r.o., Vranov N. Toplou
- South Korea (9):
  - Dong-A University Hospital, Busan
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon
  - Yeungnam Univeristy Medical Center, Gyeongsan-si
  - Inje University Haeundae Paik Hospital, Haeundae-gu
  - Kyung Hee University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University-Wonju Severance Christian Hospital, Wŏnju
- Spain (9):
  - Instituto de Ciencias Médicas, Alicante
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de GC
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital de Sagunto y C.E., Sagunto
  - Hospital Universitario Marqués de Valdecilla, Santander
- Switzerland (4):
  - Inselspital Bern, Bern
  - Gastroenterologische Praxis Balsiger, Seibold & Partner, Bern
  - Cantonal Hospital St.Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (4):
  - Antalya Egitim ve Arastırma Hastanesi, Antalya
  - Ege University Medicine of Faculty, Bornova
  - Kocaeli Üniversitesi, Kocaeli
  - Mersin University, Mersin
- Ukraine (20):
  - Communal non-profit enterprise "Regional clinical hospital of Ivano-Frankivsk Regional Council", Ivano-Frankivsk
  - City Clinical Hospital No. 2, Kharkiv
  - L.T. Mala National Institute of Therapy of NAMS of Ukraine, Kharkiv
  - Kherson City Clinical Hospital, Kherson
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kiev
  - Private Enterprise Private Manufacturing Company Acinus, Kropyvnytskyi
  - Municipal Nonprofit Enterprise of Kyiv Region Council "Kyiv Regional Clinical Hospital", Kyiv
  - Medical Center Ok!Clinic+, Kyiv
  - Municipal non-profit enterprise of Kyiv Regional Council "Kyiv Regional Center for Rehabilitation Medicine", Kyiv
  - Lviv Railway Clinical Hospital, Lviv
  - Municipal non-profit enterprise "Lviv Territorial Medical Union "Multidisciplinary Clinical Hospital of Em -T, Lviv
  - Lviv Regional Clinical Hospital - Lviv National Medical University named Danylo Galician, Lviv
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council, Odesa
  - Poltova Oblast Clinical Hospital IM.M.V.Sklifosovskoho, Poltava
  - Transcarpathian Regional Hospital im.Andriya Novak, Uzhhorod
  - City Clinical Hospital #1, Vinnitsya National Medical University, Vinnytsia
  - Medical Clinical Investigational Center of Medical Center Health Clinic, Vinnytsia
  - VNMU, Vinnytsia
  - Diaservis - Medical and Diagnostic Center, Zaporizhia
  - Diacenter, Zaporizhzhia
- United Kingdom (4):
  - Fairfield General Hospital, Bury
  - Barts Health NHS Trust, London
  - Guy's & St Thomas' NHS Foundation Trust, London
  - The John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Lilly provides access to the individual patient data from studies on approved medicines and indications as defined by the sponsor specific information on ClinicalStudyDataRequest.com.
  This access is provided in a timely fashion after the primary publication is accepted. Researchers need to have an approved research proposal submitted through ClinicalStudyDataRequest.com. Access to the data will be provided in a secure data sharing environment after signing a data sharing agreement.

REFERENCES:
- [Derived] Lee SD, Ehrlich AC, Pellanda P, Kaiser C, Todd K, Moses R, Walsh A. Long-Term Safety of Mirikizumab in Patients With Moderately to Severely Active Ulcerative Colitis: An Integrated 2-Year Safety Analysis. Am J Gastroenterol. 2025 Dec 1;120(12):2857-2866. doi: 10.14309/ajg.0000000000003407. Epub 2025 Mar 12. PMID 40071779
- [Derived] Sands BE, D'Haens G, Clemow DB, Irving PM, Johns JT, Gibble TH, Abreu MT, Lee SD, Hisamatsu T, Kobayashi T, Dubinsky MC, Vermeire S, Siegel CA, Peyrin-Biroulet L, Moses RE, Milata J, Panaccione R, Dignass A. Three-Year Efficacy and Safety of Mirikizumab Following 152 Weeks of Continuous Treatment for Ulcerative Colitis: Results From the LUCENT-3 Open-Label Extension Study. Inflamm Bowel Dis. 2025 Jul 7;31(7):1876-1890. doi: 10.1093/ibd/izae253. PMID 39448057
- See also: A Study to Evaluate the Long-Term Efficacy and Safety of Mirikizumab in Participants With Moderately to Severely Active Ulcerative Colitis (LUCENT 3) — https://trials.lillytrialguide.com/en-US/trial/3RoYr898zuoGuUiI8aiecA